CLINICAL TRIAL: NCT03743155
Title: Phase II Clinical Trial to Evaluate the Effect and Safety of MSV * in Xerostomia * Adult Autologous Bone Marrow Mesenchymal Stem Cells, Expanded Under GMP of IBGM
Brief Title: Clinical Trial to Evaluate the Effect and Safety of MSV in Xerostomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Terapia Regenerativa Tissular (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRS-ITRT-2018
Record Dates: First submitted 2018-11-05; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Xerostomia Due to Radiotherapy

STUDY DESIGN:
Intervention Model Description: single arm due to not alternative treatment exist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment with mesenchymal stem cells (Experimental): xerostomy using mesenchymal stem cells adult autologous bone marrow
  Interventions: Biological: mesenchymal cells

INTERVENTIONS:
Biological: mesenchymal cells — Autologous bone marrow aspiration is used as a cellular source to obtain MSVs and is subjected to the protocolized anticoagulant procedure. After checking the perfect condition of the shipment and the correct completion of the documentation that accompanies it, the processing of the bone marrow will be carried out. The processing of the bone marrow will be done in the Cell Therapy Unit of the IBGM under NCF, within 24 hours of the completion of the aspiration

SUMMARY:
Phase II not controlled, open-label, prospective, single center clinical trial

DETAILED DESCRIPTION:
* Determine changes in the xerostomia characteristics and discomfort degree by means of questionnaires addressed to the physician and subject of study.
* Determine the volume of submaxilar saliva without stimulation and with stimulation by sialometry (SL).
* Detect changes in volume, vascularization and fibrosis of submaxillary glands based on magnetic resonance imaging (MRI) with contrast.
* Detect changes of submaxillary gland functionalism based on Gammagraphy (GF).

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 18 to 75 years old of both sexes.
2. Biochemical analysis without significant alterations which could contraindicate the treatment.
3. Bilateral radiotherapy of the previous neck due to neoplasia in states T1-T2 and N0, N1 and N2a.
4. 2 years of follow-up without recurrence.
5. Reduction of salivation and hyposalivation, evaluated by an examination, flow rate or whole unstimulated saliva in the range of 0.05- 0.20 ml / min.
6. Grade 1-3 xerostomy as assessed by the grading scale.
7. The patient is able to understand the nature of the study.
8. Written informed consent of the patient

Exclusion Criteria:

1. Participation in another clinical trial in the 3 months prior to his/her inclusion.
2. Present infection (no infectious sign should be evidenced with repercussion on the evolution of the treated lesion).
3. Patients with positive serologies for HIV, lues and hepatitis with positive viral load.
4. History of cancer in the last 2 years. History of teratoma, adenocarcinoma derived from one of the salivary glands, lymphoma of the tonsils or some other lymphatic tissue or melanoma of pigmented cells of the oral mucosa.
5. Xerogenic medication in progress.
6. Other diseases of the salivary glands, for example, Sjögren's syndrome, sialolithiasis, etc.
7. Local infection.
8. Pregnancy or pregnancy planned within the next 2 years.
9. Breastfeeding.
10. Treatment with anticoagulants (not interruptible in MO or application).
11. Any other illness or condition that is grounds for exclusion for the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the characteristics and degree of discomfort of xerostomia trough OHIP questionnaire | 24 months
  Absolute and relative change of the score of the OHIP Questionnaire (OHIP-14-sp)
Changes in the characteristics and degree of discomfort of xerostomia. | 24 months
  Absolute and relative change of the score of the EVA Questionnaire
Sialometry results | 24 months
  Absolute and relative change in the volume of saliva (ml / min) submaxillary
Restoration of the glandular structure. | 24 months
  Changes in the glandular structure (volume) (MRI with contrast)
Restoration of the glandular structure. | 24 months
  Changes in the glandular structure (vascularization) (MRI with contrast)
Restoration of the glandular structure. | 24 months
  Changes in the glandular structure (fibrosis of submaxillary glands) (MRI with contrast)
Measurement of submaxillary gland functionalism changes based on Gammagraphy | 24 months
  Measurement of submaxillary gland functionalism changes based on Gammagraphy

SECONDARY OUTCOMES:
AEs and SAEs | 24 months
  Determination of the Safety of the proposed procedure, recording adverse events (AEs) and serious adverse events (SAEs). It will be considered as early safety measures: Pain at the site of injection, submaxillary swelling, duration of submaxillary swelling in days, oral discomfort, infection

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Terapia Regenerativa Tissular, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided